CLINICAL TRIAL: NCT02452086
Title: Effect of Low Level Laser With Ga-As (904 nm) on Expression of Angiogenic Factors (VEGF, VEGF Receptor-2,NO, HIF-1α), Oxygen Saturation of Peripheral Blood and Wound Surface Area in Ischemic Diabetic Foot Ulcers
Brief Title: Low Level Laser Therapy and Expression of VEGF, NO, VEGFR-2, HIF-1α in Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarbiat Modarres University (Other)
Responsible Party: Principal Investigator, giti torkaman, Professor of physical therapy, Physical therapy department, Faculty of medical sciences, Tarbiat modares univercity, Tarbiat Modarres University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D52.2567
Record Dates: First submitted 2015-05-10; First posted 2015-05-22 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Level Laser Therapy (Active Comparator): In laser therapy group, group who received interventions was the patients received laser with 2 Joule/centimeters2, 90 milliwatt
  , 3 days/week, for 4 weeks (12 sessions)
  Interventions: Device: Low Level Laser(Ga-As)
- Placebo (Placebo Comparator): In the placebo group, the treatment procedure was the same as that the LLLT group, but the laser light was off and Guiding light was laser was on
  Interventions: Procedure: Placebo

INTERVENTIONS:
Device: Low Level Laser(Ga-As) — Low level laser therapy(904 nm Wavelength), 90 milliwatt, 2 Joule/centimeter2
  Other Names: LLLT
  Arms: Low Level Laser Therapy
Procedure: Placebo — LLLT with zero intensity
  Other Names: Placebo low level laser therapy
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the changes of factors including Vascular Endothelial Growth Factor(VEGF), VEGFReceptor-2, Nitric Oxide and hypoxia-inducible factor-1α (HIF-1α), measurements of oxygen saturation in peripheral blood and wound surface area and ankle-brachial index (ABI) in ischemic diabetic foot ulcers after Low Level Laser Therapy(LLLT).

DETAILED DESCRIPTION:
Defects in vessels and neovascularization makes diabetic chronic wounds difficult to treat, A decrease of angiogenic factor expression such as Vascular Endothelial Growth Factor(VEGF) and its receptors is involved in angiogenesis inhibition in diabetic ulcers. LLLT as a therapeutic treatment modality can effect on release of these factors and angiogenesis in wound site.

The purpose of this study is to examine the changes of factors including VEGF, VEGFReceptor-2, Nitric Oxide and hypoxia-inducible factor-1α (HIF-1α), measurements of oxygen saturation in peripheral blood and wound surface area in ischemic diabetic foot ulcers after LLLT, Therefore, the investigators can evaluate molecular process of angiogenesis, as a mechanism of useful effects of LLLT.

In order to patients with ischemic diabetic foot ulcers(DFU) assigned into LLLT with Ga-As(904 nm) laser and placebo groups and will be treated for 12 sessions, every other day. On the first and last (twelfth) treatment session, before and after intervention, Blood sample are taken from all patients in the both groups for VEGF, VEGFreceptor-2, NO and HIF-1α measurement. Wound surface area and oxygen saturation of peripheral blood and ankle-brachial index (ABI) are measured at first and twelfth treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic diabetic foot ulcer
* Wagner classification DFU 2
* 0.5<ABI<0.9
* Mild to moderate diabetic neuropathy

Exclusion Criteria:

* Fracture in a lower limb
* A severe infection
* A malignancy
* Kidney failure
* Skin diseases
* Osteomyelitis
* Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The blood serum level of VEGF(pg/ml), VEGFR-2(pg/ml), HIF-1α(pg/ml) and NO (pg/ml) | Change from Baseline in serum level of VEGF, VEGFR-2, HIF-1α and NO at 4 weeks
  measured from serum in initial and end sessions.

SECONDARY OUTCOMES:
Wound surface area(cm2) | Change from Baseline in wound surface area at 2 and 4 weeks
Oxygen saturation of peripheral blood | Change from Baseline with pulse oximeter at 2 and 4 weeks
Ankle Brachial Index(ABI) | Change from Baselineat 2 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giti Torkaman, PHD, Study Director — Professor of Physical Therapy, Physical Therapy Department, Faculty of Medical Sciences, Tarbiat Modares Univercity
Locations (1):
- Tarbiat Modares University, Tehran, Iran

REFERENCES:
- [Derived] Torkaman G, Hoseini-Sanati M, Hedayati M, Mofid M, Iranparvar Alamdari M. Effects of Photobiomodulation Therapy on the Expression of Hypoxic Inducible Factor, Vascular Endothelial Growth Factor, and Its Specific Receptor: A Randomized Control Trial in Patients with Diabetic Foot Ulcer. Photobiomodul Photomed Laser Surg. 2024 Apr;42(4):275-284. doi: 10.1089/photob.2023.0152. Epub 2024 Mar 27. PMID 38536106